CLINICAL TRIAL: NCT04442178
Title: A Multicenter, Randomized, Double-blinded Placebo-controlled Study of Recombinant Interleukin-7 (CYT107) for Immune Restoration of Hospitalized Lymphopenic Patients With Coronavirus COVID-19 Infection. US Infectious Cohort
Brief Title: InterLeukin-7 to Improve Clinical Outcomes in Lymphopenic pAtients With COVID-19 Infection ( ILIAD-7-US-I )
Acronym: ILIAD-7-US-I
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: POOR ACCRUAL
Sponsor: Revimmune (Industry)
Collaborators: Washington University School of Medicine (Other); Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ILIAD-7 COVID US INFECTIOUS
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Lymphocytopenia
MeSH Terms: conditions — COVID-19; Lymphopenia | interventions — Interleukin-7; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: randomized controlled of treatment vs placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unblinded Pharmacist will prepare blinded syringes of colorless drug or placeb
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CYT107 Treatment (Experimental): Intramuscular (IM) administration of CYT107 twice a week for 3 weeks
  Interventions: Drug: CYT107
- Placebo (Placebo Comparator): Intramuscular (IM) administration of Saline twice a week for 3 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CYT107 — IM administration at 10μg/kg twice a week for three weeks and up to 7 administrations according to Hospital length of stay
  Other Names: Interleukin-7
  Arms: CYT107 Treatment
Drug: Placebo — IM administration at 10μg/kg twice a week for three weeks and up to 7 administrations according to Hospital length of stay
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Comparison of the effects of CYT107 vs Placebo administered IM at 10μg/kg twice a week for three weeks on immune reconstitution of lymphopenic COVID-19 patients

DETAILED DESCRIPTION:
Approximately forty-eight (48) participants will be randomized 1:1 to receive

(a) Intramuscular (IM) administration of CYT107 at 10 μg/kg followed, after 72hrs of observation, by 10 μg/kg twice a week for 3 weeks (maximum 7administrations adjusted to patient's length of stay in the hospital) or (b)Intramuscular (IM) placebo (normal saline) at the same frequency. The aim of the study is to test the ability of CYT107 to produce an immune reconstitution of these patients and observe possible association with a clinical improvement.

This cohort excludes oncology patients on treatment

ELIGIBILITY:
Inclusion Criteria:

1. A written, signed informed consent, or emergency oral consent, by the patient or the patient's legally authorized representative, and the anticipated ability for participant to be re-consented in the future for ongoing Study participation
2. Men and women aged ≥ 25 - 80 (included) years of age
3. Hospitalized patients with two absolute lymphocyte count (ALC) ≤ 1000 cells/mm3, at two time points at least 24 hours apart, following HOSPITALIZATION:
4. Hospitalized patients with moderate to severe hypoxemia requiring oxygen therapy at >4L per minute nasal cannula or greater to keep saturations >90%, non-invasive positive pressure ventilation (e.g., BIPAP), or patients intubated / ventilated for respiratory failure
5. Confirmed infection with COVID-19 by any acceptable test available / utilized at each site
6. Willingness and ability to practice contraception regardless of the gender of the patient during 5 month after last drug exposure
7. Private insurance or government / institution financial support (through CMS or other)

Exclusion Criteria:

1. Pregnancy or breast feeding
2. ALT and/or AST > 5 x ULN
3. Known, active auto-immune disease;
4. Ongoing cancer treatment with chemotherapy / immunotherapy or any cancer therapy within last 3 months and/or ongoing
5. Patients with past history of Solid Organ transplant
6. Active tuberculosis, uncontrolled active HBV or HCV infection, HIV with positive viral load
7. Hospitalized patients with refractory hypoxia, defined as inability to maintain saturation >85% with maximal available therapy for >6 hours
8. Patients receiving any agent with immune suppressive effects, other than steroids at dosages less than 300 mg/day equivalent hydrocortisone and/or anti-IL-6R treatments like Tocilizumab or Sarilumab or anti-IL-1 treatment like Anakinra which should preferably be minimized
9. Patients with baseline Rockwood Clinical Frailty Scale ≥ 6 at Hospital admission
10. Patients showing an increase of the NEWS2 score by more than 6 points during the screening/ baseline period (48 to 72 hrs prior to first administration)
11. Patients under guardianship

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Improvement of the absolute lymphocyte count (ALC) of lymphopenic (ALC≤1000/mm3) COVID-19 infected participants out to approximately 30 days following initial Study drug administration or Hospital discharge (HD), whichever occurs first | one month
  A statistically significant increase of the absolute lymphocyte count (ALC) from randomization to day 30 or Hospital Discharge

SECONDARY OUTCOMES:
To obtain "clinical improvement" as defined by an improvement in a 11-points WHO score for Clinical Assessment, through day 30 or HD. | one month
  to determine if CYT107 will improve the clinical status of hospitalized COVID-19 patients as measured by 11 steps WHO clinical improvement score
a significant decline of SARS-CoV-2 viral load through day 30 or HD | one month
  The decrease of SARS-CoV-2 viral load from measurements at baseline and days of treatment dose 4 and dose 5, Day 21 and Day 30 or HD (whichever occurs first)
frequency of secondary infections through day 45 compared to placebo arm | 45 days
  Incidence of secondary infections based on pre-specified criteria as adjudicated by the Secondary Infections Committee (SIC) through Day 45
length of hospitalization compared to placebo arm | 45 days
  Number of days of hospitalization during index hospitalization (defined as time from initial Study drug treatment through HD)
Length of stay in ICU compared to placebo arm | 45 days
  Number of days in ICU during index hospitalization
number of readmissions to ICU compared to placebo arm | 45 days
  Readmissions to ICU through Day 45
organ support free days compared to placebo arm | 45 days
  Organ support free days (OSFDs) during index hospitalization (This includes ventilator assistance free days)
Frequency of re-hospitalization through day 45 compared to placebo arm | 45 days
  Number of readmissions to the hospital through Day 45
All-cause mortality through day 45 compared to placebo arm | 45 days
  All-cause mortality through Day 45
CD4+ and CD8+ T cell counts compared to placebo arm | 30 days
  Absolute numbers of CD4+ and CD8+ T-cell counts at time points indicated on the Schedule of Activities (SoA)through Day 30 or HD
level of other known biomarkers of inflammation: Ferritin compared to placebo a | 30 days
  Track and evaluate other known biomarkers of inflammation, Ferritin, from baseline to day 30
Level of other known biomarkers of inflammation: CRP compared to placebo arm | 30 days
  Level of other known biomarkers of inflammation: CRP compared to placebo arm
Level of other known biomarkers of inflammation: D-dimer compared to placebo arm | 30 days
  Track and evaluate other known biomarkers of inflammation, D-dimer from baseline to day 30
Physiological status through NEWS2 evaluation compared to Placebo arm | 30 days
  Evaluate improvement of the NEWS2 score value. Score form 0 to 4: NO Risk Score of 7 or more: High risk

OTHER OUTCOMES:
Safety assessment through incidence and scoring of grade 3-4 adverse events | 45 days
  Incidence and scoring of all grade 3-4 adverse events through Day 45 (using CTCAE Version 5.0) to assess safety

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hotchkiss, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (5):
  - University of Florida College of Medicine, Gainesville, Florida
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Rutgers Health, New Brunswick, New Jersey
  - Stony Brook Medicine, Stony Brook, New York
  - Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
Publication

REFERENCES:
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Francois B, Jeannet R, Daix T, Walton AH, Shotwell MS, Unsinger J, Monneret G, Rimmele T, Blood T, Morre M, Gregoire A, Mayo GA, Blood J, Durum SK, Sherwood ER, Hotchkiss RS. Interleukin-7 restores lymphocytes in septic shock: the IRIS-7 randomized clinical trial. JCI Insight. 2018 Mar 8;3(5):e98960. doi: 10.1172/jci.insight.98960. PMID 29515037
- [Result] Venet F, Foray AP, Villars-Mechin A, Malcus C, Poitevin-Later F, Lepape A, Monneret G. IL-7 restores lymphocyte functions in septic patients. J Immunol. 2012 Nov 15;189(10):5073-81. doi: 10.4049/jimmunol.1202062. Epub 2012 Oct 10. PMID 23053510
- [Derived] Shankar-Hari M, Francois B, Remy KE, Gutierrez C, Pastores S, Daix T, Jeannet R, Blood J, Walton AH, Salomao R, Auzinger G, Striker D, Martin RS, Anand NJ, Bosanquet J, Blood T, Brakenridge S, Moldawer LL, Vachharajani V, Yee C, Dal-Pizzol F, Morre M, Berbille F, van den Brink M, Hotchkiss R. A randomized, double-blind, placebo-controlled trial of IL-7 in critically ill patients with COVID-19. JCI Insight. 2025 Feb 4;10(6):e189150. doi: 10.1172/jci.insight.189150. PMID 39903535